## **Statistical Analysis Plan**

# THRIVE (Tradespeople and Hand-workers Rural Initiative for a Vision-enhanced Economy) randomized controlled trial

### Reading Glasses on Livelihoods and Quality of Life in Rural Bangladesh

ClinicalTrials.gov identifier: NCT03719196

#### **DOCUMENT HISTORY**

| Version | Date | Edited by | Comments | Timing in relation to unblinding |
|---|---|---|---|---|
| 2.0 | March 2021 | NC | | |

#### **CONTRIBUTORS**

Nathan Congdon (QUB), Susan Bergson (VisionSpring)

#### **ANALYSIS**

#### 1. Analysis of primary and secondary outcomes

Differences in baseline characteristics by study group will be analysed using the t-test or Wilcoxon rank-sum test for continuous variables with or without normal distribution respectively, the Chi-squared or Fisher's exact test (with cell frequency<5) for binary categorical variables, and ordinal logistic regression for ordinal categorical variables. Normality will be checked using histograms and Q-Q plots.

Data for the primary outcome will be presented as median and inter quartile range due to lack of normality, the change in self-reported monthly income will be categorized by quartiles and the unadjusted and adjusted intervention effects, odds ratio and 95% CI estimated using ordinal logistic regression. Unadjusted and adjusted mean between-group differences will be estimated for the secondary outcomes using linear regression. All variables with P<0.05 in the simple regression analysis will be included in multiple regression models. All statistical analyses will be performed using a commercially available software package (Stata 15.1, StataCorp, College Station TX, USA).